CLINICAL TRIAL: NCT06849700
Title: Can Active Gamification Improve the Physical and Mental Health of Primary School Children?
Brief Title: Effects of Active Gamification in Primary School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: *University of Jaén*
Record Dates: First submitted 2025-02-17; First posted 2025-02-27 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Students; Mental Health Issue; Physical Condition

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group continued with their traditional Physical Education classes.
- Experimental Group (Experimental): The experimental group participated in a program based on the gamification of physical exercise
  Interventions: Other: Active gamification

INTERVENTIONS:
Other: Active gamification — The experimental group participated in a physical exercise program for primary school children, with 45-minute sessions three times a week, including warm-up, main activities, and awards. Designed to enhance engagement through game mechanics, the program progressed in three phases: Explorers in Action (Weeks 1-4) focused on coordination, agility, and teamwork with games like "Conquering Territories"; Movement Heroes (Weeks 5-8) emphasized endurance, collaboration, and strategy through activities like "Quest for the Gems"; and Health Guardians (Weeks 9-12) incorporated strength, planning, and teamwork challenges, culminating in a final integrated skills circuit. The program promoted continuous improvement in physical and cooperative abilities.
  Arms: Experimental Group

SUMMARY:
Active gamification, which incorporates game elements with physical interaction, is presented as an innovative strategy to address children's physical and mental health. This study aims to evaluate the impact of an active gamification program on these variables in primary school children. To this end, a randomized clinical trial will be conducted with 120 children between the ages of 8 and 11. Participants will be randomly assigned to one of two groups: an experimental group, which will participate in a program designed to promote physical activity through game-based dynamics for 12 weeks, and a control group, which will continue with traditional physical education classes without modifications to their usual methodology. The program implementation includes structured sessions with activities designed to encourage interaction, movement, and decision-making in a playful environment, with the aim of improving children's engagement and adherence to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age between 8 and 11 years
* No medical contraindication for physical activity
* No intellectual disability that could interfere with understanding or compliance with the study procedures; and iv) informed consent from parents or legal guardians.

Those students who did not meet the inclusion criteria were able to participate in the intervention with their peers, but were not considered in the analysis.

Exclusion Criteria:

* Diagnosis of neuromotor disorder or severe physical disability that limits participation in the scheduled physical activity
* Presence of severe psychological or behavioral disorders that make integration into group activities difficult.
* Use of medication that significantly affects physical or cognitive performance.
* Failure to attend more than 20% of the intervention program sessions
* Withdrawal of informed consent by parents or legal guardians during the study

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2024-10-08 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
Anxiety | Up to twelve weeks
  Anxiety will be assessed using the short version of the Spence Children's Anxiety Scale for Spanish children (SCAS-C-8), in its version validated in Spanish. This scale consists of 18 items, each of them rated on a Likert-type scale from 0 to 3 (0 = Never, 1 = Sometimes, 2 = Often and 3 = Always), where higher scores indicate a greater presence of anxiety symptoms.
Sleep quality | Up to twelve weeks
  The Children's Sleep Habits Questionnaire (CSHQ) assesses sleep quality in children using 33 items rated on a Likert scale (1-3), with total scores ranging from 33 to 99, where higher scores indicate more sleep problems. The Spanish-validated version was used in this study. The questionnaire is divided into eight subscales: Bedtime Resistance, Sleep Onset Delay, Sleep Duration, Sleep Anxiety, Night Wakings, Parasomnias, Sleep-Disordered Breathing, and Daytime Sleepiness. The CSHQ Global Score is the sum of all items.
Self-Esteem | Up to twelve weeks
  The self-esteem test for schoolchildren, in its Spanish version, evaluates how the student perceives themselves through 25 items, of which 23 are statements that are answered with either "YES" or "NO." Scoring is done using a template provided by the author, where the correct answers for a high self-esteem level are indicated. If the student's answer matches the template, 1 point is awarded; if it does not, no points are given. The items with "NO" answers are 1, 4, 8, 10, 12, 13, 15, 16, 17, 19, 20, and 21, while the "YES" answers are 2, 3, 5, 6, 7, 9, 11, 14, 18, 22, and 23. Based on the total score (PD), the self-esteem level is determined: 22-25 points, high self-esteem; 17-21 points, tendency toward high self-esteem; 16 points, at-risk self-esteem; 12-15 points, tendency toward low self-esteem; and 11 or fewer points, low self-esteem.
Self-Concept | Up to twelve weeks
  The Garley Self-Concept Questionnaire, validated in Spanish for primary school students, consists of 48 statements divided into six dimensions: (a) physical self-concept, (b) social acceptance, (c) family self-concept, (d) intellectual self-concept, (e) personal self-evaluation, and (f) sense of control. Each dimension has 8 items. Responses are measured on a 5-point Likert scale: never (1), rarely (2), I could not say (3), often (4), and always (5). The questionnaire includes both direct (items 1-2, 4-7, 9-10, etc.) and inverse (items 3, 8, 11, etc.) items. For direct items, scoring follows the standard scale, while for inverse items, the scale is reversed. The scores for each subscale range from 8 to 40 points, with higher scores indicating a better self-concept. The overall score is calculated by summing the individual items.
Social Skills | Up to twelve weeks
  The Matson Evaluation of Social Skills in Youngsters (MESSY), in its Spanish version, was used to assess social skills in students. The questionnaire includes a four-step response format: never, sometimes, often, and always. It evaluates five factors: appropriate social skills (24 items) such as making friends and emotional expressiveness (e.g., "I look at people when I talk to them"); inappropriate assertiveness (16 items) addressing aggressive behaviors (e.g., "I take things that are not mine without permission"); impulsivity (5 items) such as getting easily angry (e.g., "I interrupt others when they are speaking"); overconfidence (6 items) involving self-overvaluation (e.g., "I like to brag to others about the things I have"); and jealousy/loneliness (4 items) exploring feelings of isolation (e.g., "I feel lonely"). Only the student version of MESSY was used in this study.
Concentration and Selective Attention | Up to twelve weeks
  The D2 test, in its Spanish version, assesses selective attention and concentration in the school context. The participant's task is to carefully check, starting from left to right, what is written on each line and must mark all the letters that have two small lines (two lower, two upper, or one lower and one upper) with a "d". These elements are considered relevant. The other combinations (the "d" and the "p", with and without lines) are known as irrelevant, and should not be marked. The participant has 20 s for each line. This test has demonstrated excellent reliability, with ranges between 0.90 and 0.97 for both Cronbach's α and the test-retest, and has also shown convergent and divergent validity.
Creativity | Up to twelve weeks
  The Creative Intelligence Test (CREA) is used to assess creative intelligence by cognitively assessing creativity on an individual basis by reproducing question indicators within a theoretical context of research and problem solving. The procedure consists of showing a photograph to the child and asking him to fill in the blank spaces at the top of the copy with the data that appear. The task is based on writing, briefly, as many pre-questions as possible about what it shows. The CREA test has been found to meet the standards of reliability and validity required for a psychological test (Cronbach's α = 0.875).
Memory | Up to twelve weeks
  To assess memory, a 1-minute ad hoc test was used, based on the original ideas of the memory test included in the Spanish adaptation of the Reynolds Intelligence Scale [RIAS]. A poster of 15 randomly selected Spanish playing cards was projected for 20 seconds on a 3 x 2 meter screen. Immediately afterward, participants had 40 seconds to record on a standardized sheet the greatest number of cards they could remember. The total number of correct answers was counted (range 0-15). Before the test, it was verified that all participants knew the structure and content of the 40 cards in the Spanish deck.
Aerobic capacity | Up to twelve weeks
  This will be determined using the 20-meter Course Navette Test, an incremental test in which participants must run from end to end over a distance of 20 meters, following an audible signal and increasing their speed in 0.5 km/h intervals every minute. The test will begin at a speed of 8.5 km/h and will end when the participant fails to maintain the pace on two consecutive attempts or stops. In each case, the number of periods passed will be recorded at the end of the test. This test will be administered only once at the end of the data collection session.
Speed and agility | Up to twelve weeks
  The 4x10-meter shuttle test will be used, in which students must cover the distance four times at maximum speed.
Muscular strength | Up to twelve weeks
  This will be measured through three tests: i) upper body strength will be assessed using a handheld dynamometer, in which a handheld dynamometer will be used for each limb; ii) lower body strength will be analyzed using the horizontal jump test without momentum; and iii) a muscular endurance test will also be performed with a 30-second sit-up test.
Flexibility | Up to twelve weeks
  This test will be assessed using the Sit-and-Reach test. The test will be performed using a special 33 cm box with a sliding ruler attached to the top. Participants will sit on the floor with their knees extended, shoulder-width apart, and their feet in contact with the bottom of the box. They will be asked to bend their torso and extend their arms forward as far as possible, holding the final position for at least two seconds. The test will be performed twice, and the best result in centimeters will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Agustín Aibar Almazán, Jaén, Spain